CLINICAL TRIAL: NCT01335438
Title: Total Knee Arthroplasty Comparing Cementless to Cemented Fixation, A Prospective Comparison of Long Term Outcomes Using and Identical Design of Prosthesis
Brief Title: Total Knee Arthroplasty Comparing Cementless to Cemented Fixation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Young Hoo Kim (Other)
Responsible Party: Sponsor-Investigator, Young Hoo Kim, Professor and Director, Ewha Womans University
Organization: Ewha Womans University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TKRcementless
Record Dates: First submitted 2011-04-11; First posted 2011-04-14 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Osteoarthritis
Keywords: total knee arthroplasty; cemented; cementless; fixation; posterior stabilized; cruciate retaining
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cementless Nexgen CR (Experimental): Cementless fixation of Nexgen CR TKR
  Interventions: Device: Cementless (Nexgen)
- Cemented Nexgen CR (Active Comparator): Cemented fixation of Nexgen CR TKR
  Interventions: Device: Cemented (Nexgen)

INTERVENTIONS:
Device: Cementless (Nexgen) — Cementless fixation of Nexgen CR TKR
  Other Names: Cementless Nexgen
  Arms: Cementless Nexgen CR
Device: Cemented (Nexgen) — Cemented fixation of Nexgen CR TKR
  Other Names: Cemented Nexgen
  Arms: Cemented Nexgen CR

SUMMARY:
The purpose of this study is to determine if there are any clinical or radiographic differences in cemented and cementless fixation in total knee replacement.

DETAILED DESCRIPTION:
Out comes measures were to determine:

1. whether the knee and function scores and the radiographic results of the knees with a Nexgen cemented knee prosthesis would be better than those with an Nexgen cementless prosthesis.
2. whether the patients with a Nexgen cemented knee prosthesis would have a better range of knee motion than those with an Nexgen cementless prosthesis.
3. whether patient satisfaction and preference would be better in the patients having a Nexgen cemented knee prosthesis than those of patients having an Nexgen cementless knee prosthesis
4. whether complication rate would be less in the knees with a Nexgen cemented knee prosthesis than in the knees with an Nexgen cementless prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* End-stage osteoarthritis of the knee joint requiring total knee arthroplasty with bilateral disease

Exclusion Criteria:

* Inflammatory disease
* patient with other Lower extremity disease which may affect functional outcome
* Neurologic disease effecting patients lower extremity
* Revision surgery
* Patient not medically cleared for bilateral surgery

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 1997-01; Primary Completion 1998-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Improvement in Knee Society Knee Score | Initial(one day before surgery), and at 3 months, 1 year, then annually after surgery
  change in knee score will be compared with initial score, until mean follow up of 25 years.

SECONDARY OUTCOMES:
Improvement in the Range of Motion | Initial(one day before surgery), and at 3 months, 1 year, then annually after surgery
  change in the range of motion of knee joint will be compared with the initial value, until mean follow up of 25 years.

CONTACTS AND LOCATIONS:
Overall Officials: Jang Won Park, MD, Principal Investigator — Ewha Womans University Mokdong Hospital
Locations (1):
- Ewha Womans University Mokdong Hosptial, Seoul, South Korea